CLINICAL TRIAL: NCT05313906
Title: Disitamab Vedotin Plus Penpulimab and Cisplatin in Advanced Gastric Cancer
Brief Title: RC48 Plus AK105 and Cisplatin in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Rongchang Biopharmaceutical (Unknown); Zhengda Tianqing Pharmaceutical Group Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Quanli Gao, Dr, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH immunotherapy007
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Advanced Gastric Carcinoma; HER2-positive Gastric Cancer

STUDY DESIGN:
Intervention Model Description: RC48 plus AK105 and cisplatin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exprimental group (Experimental): RC48 plus AK105 and cisplatin
  Interventions: Drug: RC48+AK105+cisplatin

INTERVENTIONS:
Drug: RC48+AK105+cisplatin — RC48 plus AK105 and cisplatin

SUMMARY:
To explore the safety and clinical efficacy of cisplatin combined with RC48 and anti-PD-1 antibodies AK105 in Her-2 positive advanced gastric cancer.

DETAILED DESCRIPTION:
Although anti-PD-1 antibody could prolong the survival of patients with adanced gastic cancer, there are relatively few reports on anti-PD-1 antibody therapy in Her2-positive gastric cancer. RC48 is a primary anti-HER2 antibody-drug conjugate, which has been approved by the Chinese NMPA for the later-line treatment of Her2-positive gastric cancer. This study was to explore the safety and clinical efficacy of RC48 combined with cisplatin and AK105 in previously untreated patients with HER2-positive gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, ≤75 years old, regardless gender
* Pathologically confirmed gastric adenocarcinoma, Her2 immunohistochemical examination of 2+ or 3+
* ECOG PS scores 0-1
* Stage IV according to AJCC 8.0 and no systemic therapy previously
* Expected lifespan ≥ 3 months
* Adequate organ function
* At least one measurable lesion according to RECIST 1.1
* Asymptomatic intracranial metastasis
* No history of other malignancies
* Women of childbearing age must have a negative blood pregnancy test within 7 days, and subjects of childbearing age must use appropriate contraception during the trial and for 6 months after the trial
* Agreed to participate in this clinical study and signed the Informed Consent

Exclusion Criteria:

* Currently participating in an interventional clinical investigational treatment, or have received other investigational drugs or treatment with an investigational device within 4 weeks prior to the first dose
* Received anti-PD-1, anti-PD-L1, anti-CTLA-4, and other checkpoint inhibitor
* Received traditional Chinese medicines or immunomodulatory drugs with anti-gastric cancer indications within 2 weeks before the first administration
* Active autoimmune diseases or immunodeficiency diseases
* Allergy to any test drug and its excipients, or a history of severe allergy, or contraindication to the test drug
* Severe mental disorder
* Receiving systemic corticosteroids within 7 days prior to the first dose of the study
* Clinically apparent cardiovascular and cerebrovascular disease
* Others investigators evaluated not meet the inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-07 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
ORR | three months
  the proportion of patients who got CR and PR

SECONDARY OUTCOMES:
PFS | six months and twelve months
  the duration of diseases stable or better
DCR | three months
  the proportion of patients who got CR, PR and SD

CONTACTS AND LOCATIONS:
Overall Officials: Quanli Gao, Dr, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: The IPD will be shared with researhers who plan to do meta-analysis or other reasonable requests.